CLINICAL TRIAL: NCT01821547
Title: Hepatitis B Immunisation: A Two-part Study Investigating Antigen Specific B Cell Receptors
Brief Title: New Methods to Measure the Immune Response to Hepatitis B Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OVG 2012/09
Record Dates: First submitted 2013-03-18; First posted 2013-04-01 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2016-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hepatitis B vaccine — Immunisation with HepB vaccine (HBvaxPRO, 10μg/ml, Sanofi Pastuer) via intramuscular injection into the non-dominant deltoid (part 1 only).
  Other Names: HBvaxPRO, 10μg/ml, Sanofi Pastuer

SUMMARY:
Hepatitis B vaccine is a safe and effective vaccine used widely throughout the world. Because of this it is a useful vaccine in which to develop new methods for studying immune responses. Measuring the immune response to vaccines helps us to understand how they work and whether they are likely to protect any individual against infection. For most vaccines we measure the immune system's production of antibody after a vaccine has been given. The investigators want to develop new methods that give a far more detailed picture of the antibody response to vaccines than has previously been possible. These methods will investigate the genetic instructions used by each antibody producing cell to make antibody. These methods have the potential to give new insights into the way vaccines work, which could be applied to studying vaccines and vaccine schedules in the future.

ELIGIBILITY:
Inclusion Criteria:

All participants for both parts 1 and 2 must meet the following conditions in order to be enrolled:

* Participant is willing and able to give informed consent for participation in the study
* Healthy Male or Female, aged 18 - 60 years
* No allergies to the vaccine or its excipients

Participants enrolling in Part 1 must also meet the following conditions:

* Participant has previously received a primary immunisation course of HepB vaccine (3 primary doses). The 4th booster dose recommended after 12 months is not a requirement. There are a variety of possible recommended schedules, and any may have been used as long as the final vaccine (or booster vaccine) was given at least 12 months prior to the participant enrolling in the study.
* Participant is willing to allow their General Practitioner to be notified, if appropriate, of participation in the study

Participants enrolling in Part 2 must also meet the following conditions Participant receiving HBvaxPro® (the usual vaccine given within the Occupational Health Department).

Exclusion Criteria:

The participant may not enter either study if ANY of the following apply:

* Have any known or suspected impairment or alteration of immune function, resulting from, for example:

  * Congenital or acquired immunodeficiency (including IgA deficiency)
  * Human Immunodeficiency Virus infection or symptoms/signs suggestive of an HIV-associated condition
  * Autoimmune disease
  * Receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 12 months or long-term systemic corticosteroid therapy.
  * Chronic illness that could interfere with immunological function or donation of the required volumes of blood (e.g. cardiac or renal disease, diabetes, or auto-immune disorders).
* Receipt of a HepB booster vaccine within the past 12 months.
* Prior history of anaphylactic reaction to a previous dose of a Hepatitis B containing vaccine or known hypersensitivity to any vaccine component;
* Receipt of blood, blood products, or plasma derivatives within the past 3 months.
* Total blood donation greater than 50 ml within the past 3 months.
* Thrombocytopenia or any bleeding disorder.
* Pregnancy as confirmed by a positive pregnancy test, or currently breastfeeding.
* Receipt of a live vaccine within 4 weeks prior to vaccination or a killed vaccine within 7 days prior to vaccination.
* Plan to receive any vaccine other than the study vaccine within 4 weeks following vaccination.
* Enrolled in another study, which, in the opinion of the investigator, could compromise the integrity of either study being conducted.
* A member of staff on the delegation log
* According to the TOPS database, have recently taken part in a significant number of other studies, which, in the opinion of the investigator, warrant exclusion from further studies.
* Participant is a known non-responder to the HepB vaccine
* Have any condition, which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* Unable to understand English, or what will be required from them during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Part 2- To assess B cell VH/L gene segment usage by HepB specific B cells during and following administration of a three dose course of HepB vaccine given at 0,1, 2 or 0, 1, 6 months. | 0 and 7 days after the second immunisation, and 0, 7 and 40 days after the third immunisation
  HepB specific cells will be isolated using magnetic-activated cell sorting, and fluorescence-activated cell sorting. VH/L gene segments will be amplified by PCR, and DNA prepared for sequencing. Bioinformatic approaches will then be used to create frequency tables of the different V, D and J exons that comprise these gene segments.
Part 1- To validate B cell assays and assess the kinetics of HepB specific B cell subsets following administration of a booster dose of HepB vaccine given to previously immunised healthy adults. | 0, 7, 14, 21 and 28 days after immunisation
  HepB specific B cell subsets will be identified using both ELISPOT and flow cytometry.

SECONDARY OUTCOMES:
Part 1 • To measure HepB surface antigen-specific antibody concentration following administration of a booster dose of HepB vaccine given to previously immunised healthy adults | 0 and 28 days after immunisation
  Antibody concentrations will be determined from blood plasma using an ELISA
Part 1 • To assess B-cell receptor VH/L gene sequences used in HepB specific and non-antigen specific B-cells prior to and following administration of a booster dose of HepB vaccine given to previously immunised healthy adults | 0, 7, 14, 21 and 28 days after immunisation
  VH/L gene segments will be amplified by PCR, and DNA prepared for sequencing. Bioinformatic approaches will then be used to create frequency tables of the different V, D and J exons that comprise these gene segments.
Part 1 • Comparison of B cell receptor VH/L gene segment usage as determined by two different next-generation sequencing methods (RNA-sequencing and 454). | 0, 7, 14, 21 and 28 days after immunisation, as required
  Different sequencing protocols introduce different types of error and bias into the resulting sequence datasets. VH/L gene segments will sequenced using two different techniques. Bioinformatic approaches and descriptive analysis will then be used to compare the effects of the two different protocols. Frequency tables of the different V, D and J exons that comprise these gene segments will be generated, for comparison.
Part 1 • Collection of mRNA for subsequent gene expression analysis | 0, 7, 14, 21 and 28 days after immunisation
Part 2 • To measure HepB specific plasma and memory B cell frequencies during and following administration of a three dose course of HepB vaccine given at 0, 1, 2 or 0, 1, 6 months. | 0 and 7 days after the second immunisation, and 0, 7 and 40 days after the third immunisation
  HepB specific B cell subsets will be identified using both ELISPOT and flow cytometry.
Part 2 • To measure HepB surface antigen-specific antibody concentration during and following administration of a three dose course of HepB vaccine given at 0,1, 2 or 0, 1, 6 months. | 0 days after the second immunisation, and 0 and 40 days after the third immunisation
  Antibody concentrations will be determined from blood plasma using an ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Kelly, Principal Investigator — Oxford Vaccine Group
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom